CLINICAL TRIAL: NCT03223454
Title: Safety and Therapeutic Effect of Human Amniotic Epithelial Cells in Severe Refractory Asherman's Syndrome
Brief Title: Human Amniotic Epithelial Cells for Asherman's Syndrome
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Collaborators: Shanghai iCELL Biotechnology Co., Ltd, Shanghai, China (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-116
Record Dates: First submitted 2017-07-13; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Asherman's Syndrome
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- biological amnion loaded with hAECs (Experimental): Biological amnion loaded with 100 million hAECs is placed into uterine cavity immediately after TCRA.
  Interventions: Biological: hAECs
- biological amnion (Placebo Comparator): Biological amnion is placed into uterine cavity immediately after TCRA.
  Interventions: Biological: biological amnion
- intravenous infusion of hAECs (Experimental): intravenous infusion of 100 million hAECs immediately after TCRA
  Interventions: Biological: hAECs
- intrauterine infusion of hAECs (Experimental): 100 million hAECs is infused into uterine cavity immediately after TCRA.
  Interventions: Biological: hAECs
- hydrogel loaded with hAECs (Experimental): Hydrogel loaded with 100 million hAECs is infused into uterine cavity immediately after TCRA.
  Interventions: Biological: hAECs

INTERVENTIONS:
Biological: hAECs — hAECs are provided by Chongqing iCELL Biotechnology Co.,Ltd., which is a subsidiary of Shanghai iCELL Biotechnology Co.,Ltd. The participants are blind to their arms because the surgery is done under anesthesia. After hysteroscopic adhesiolysis, subsequently oral antibiotics will be given for 3 days to prevent infection. Estrogen will be administrated for 3 cycles to stimulate the repair of endometrium after the surgery.
  Arms: biological amnion loaded with hAECs; hydrogel loaded with hAECs; intrauterine infusion of hAECs; intravenous infusion of hAECs
Biological: biological amnion — Biological amnion is purchased from JiangXi RuiJi BioTechnology Co.,Ltd. The participants are blind to their arms because the surgery is done under anesthesia. After hysteroscopic adhesiolysis, subsequently oral antibiotics will be given for 3 days to prevent infection. Estrogen will be administrated for 3 cycles to stimulate the repair of endometrium after the surgery.
  Arms: biological amnion

SUMMARY:
This project aims to investigate the safety and effectiveness of human amniotic epithelial cells in the treatment of the severe refractory Asherman's syndrome.

DETAILED DESCRIPTION:
Asherman's syndrome is a gynecological disorder caused by the destruction of the endometrium due to repeated or aggressive curettages and/or endometritis. As a result, there is a loss of functional endometrium in multiple areas and the uterine cavity is obliterated by intrauterine adhesions, which results in amenorrhea, hypomenorrhea, infertility and recurrent pregnancy loss. Transcervical resection of adhesion (TCRA) is the main treatment for Asherman's syndrome, so far the effect is usually poor in moderate to severe refractory cases.

Human amniotic epithelial cells (hAECs) are derived from human amniotic epithelium. hAECs retain the characteristics approximating to embryonic stem cells. Animal experiments have shown that the endometrial thickness and fertility of mice were significantly improved after intrauterine therapy with amniotic epithelial cells. To further explore the role of hAECs in Asherman's syndrome patients, this project plans to evaluate the safety of hAECs provided by Chongqing iCELL Biotechnology Co.,Ltd., which is a subsidiary of Shanghai iCELL Biotechnology Co.,Ltd., and find an effective treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

* 1. Hysteroscopy examination confirms intrauterine adhesions, II -III according to the American Fertility Society (AFS) classification of uterine adhesions;
* 2. Regular Menstrual cycles and menstruation is normal before abortion or curettage;
* 3. Having a clear desire to fertility;
* 4. Normal blood coagulation, liver, heart, and kidney function, absence of HIV, Hepatitis B or C, syphilis and psychiatric pathology;
* 5. Serum β-hCG is negative;
* 6. Be willing to complete the study and sign the consent form.

Exclusion Criteria:

* 1. Having a history of malignant tumor;
* 2. Having other uterine diseases, such as, uterine fibroids, adenomyosis and uterine malformations;
* 3. Hysteroscopic adhesiolysis more than 3 times in the past;
* 4. Absence of peripheral vein access.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Menstrual blood volume | at 3 months
  Estimate the menstrual blood volume after surgery by the number of sanitary napkins per day and number of days, which will be compared with pre-operation.

SECONDARY OUTCOMES:
Endometrial thickness | at 3 months
  Measure the endometrial thickness during periovulatory period on ultrasound by the same trained medical sonographers at 3 months after surgery, compared with pre-operation.
Uterine volume | at 3 months
  Measure the uterine volume during periovulatory period on ultrasound by the same trained medical sonographers at 3 months after surgery, compared with pre-operation.
Ongoing pregnancy rate | up to 24 months
  A ongoing pregnancy means that at the 12th week of pregnancy, ultrasound reveals that the fetus had a heart beat and the size of the fetus is in consistent with the gestational week.

CONTACTS AND LOCATIONS:
Overall Officials: Lina Hu, Study Chair — The Second Affiliated Hospital of Chongqing Medical University; Chanyu Zhang, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University; Fan He, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University; Jianguo Hu, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University; Heng Zou, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University; Huijia Chen, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University

REFERENCES:
- [Background] Yu D, Wong YM, Cheong Y, Xia E, Li TC. Asherman syndrome--one century later. Fertil Steril. 2008 Apr;89(4):759-79. doi: 10.1016/j.fertnstert.2008.02.096. PMID 18406834
- [Background] Ilancheran S, Moodley Y, Manuelpillai U. Human fetal membranes: a source of stem cells for tissue regeneration and repair? Placenta. 2009 Jan;30(1):2-10. doi: 10.1016/j.placenta.2008.09.009. Epub 2008 Nov 7. PMID 18995896